CLINICAL TRIAL: NCT00200044
Title: Gatekeeper® System Sham-Controlled Study for the Treatment of GERD
Brief Title: An Evaluation of the Medtronic Gatekeeper System in the Treatment of SUBJECTS With Gastroesophageal Reflux Disease (GERD)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of efficacy
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Chad Giese / Clinical Research Specialist, Medtronic Neuromodulation - Gastroenterology and Urology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MGU - 002
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sham (Sham Comparator): This arm of the study has the procedure but does not get the Gatekeeper prostheses. The Sham arm has the option to cross-over to the Treatment arm at the 6-month visit.
  Interventions: Device: Gatekeeper Reflux Repair System
- Treatment (Active Comparator): The treatment arm has the Gatekeeper devices implanted.
  Interventions: Device: Gatekeeper Reflux Repair System

INTERVENTIONS:
Device: Gatekeeper Reflux Repair System — The Gatekeeper System™ consists of a specialized 16-mm overtube assembly, a 2.4-mm diameter prosthesis delivery system (1-mm diameter needle, dilator, and 2.4-mm diameter sheath), a pushrod assembly and Gatekeeper Prosthesis. Up to 4 prostheses will be implanted at the initial procedure and retreatment with up to four more prostheses will be allowed at 3-months if the subject has a GERD HRQL score >15.
  Other Names: Gatekeeper

SUMMARY:
The purpose of the study is to demonstrate the intended use of the Gatekeeper Reflux Repair System to provide symptomatic relief is subjects with gastroesophageal reflux disease.

DETAILED DESCRIPTION:
The purpose of the study is to demonstrate the intended use of the Gatekeeper Reflux Repair System to provide symptomatic relief is subjects with gastroesophageal reflux disease

ELIGIBILITY:
Diagnosis and main criteria for inclusion:

* Subjects diagnosed with GERD with symptomatic improvement on PPIs.
* Subjects who have demonstrated a baseline 24 Hour pH ≥ 4% time with pH ≤ 4.0.
* Subjects with a baseline GERD-HRQL heartburn score of ≤11 on PPI and ≥ 20 off PPI.

Diagnosis and main criteria for exclusion:

* Extensive Barrett's Esophagus (> 2 cm).
* Esophagitis (LA Classification Grades C or D).
* Previous history of gastroesophageal surgery, anti-reflux procedures, or gastroesophageal or gastric cancer.
* Large hiatal hernia (> 3 cm).
* Current complaints of clinical dysphagia evidenced by greater than one occurrence per month.
* Esophageal strictures
* Esophageal or gastric varices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2002-12; Primary Completion 2006-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Reduction in serious device and procedure related adverse device effects. | 6 months

SECONDARY OUTCOMES:
Improvement in espophageal pH | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Glen Lehman, Principal Investigator — Indiana University Hospital
Locations (11):
- United States (10):
  - Contact Medtronic for specific site information, San Francisco, California
  - Contact Medtronic for specific site information, Atlanta, Georgia
  - Contact Medtronic for specific site information, Chicago, Illinois
  - Contact Medtronic for specific site information, Indianapolis, Indiana
  - Contact Medtronic for specific site information, Lexington, Kentucky
  - Contact Medtronic for specific site information, St Louis, Missouri
  - Contact Medtronic for specific site information, Lebanon, New Hampshire
  - Contact Medtronic for specific site information, New York, New York
  - Contact Medtronic for specific site information, Knoxville, Tennessee
  - Contact Medtronic for specific site information, Milwaukee, Wisconsin
- Contact Medtronic for specific site information, Amsterdam, Netherlands